CLINICAL TRIAL: NCT01296152
Title: An Open-Label, Non-Randomized Study of Pharmacokinetic Interactions Between Depo-Medroxyprogesterone Acetate (DMPA) and Lopinavir/Ritonavir (LPV/r) and of the Effects of DMPA on Cellular Immunity and Regulation in HIV-Infected Women
Brief Title: Pharmacokinetic Interactions Between DMPA and LPV/r Among HIV-Infected Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5283; 1U01AI068636 (NIH)
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-11

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Medroxyprogesterone Acetate; N,N-dimethyl-4-anisidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Depo-medroxyprogesterone acetate (DMPA) (Experimental): At study entry/ Day 0, subjects will receive depo-medroxyprogesterone (DMPA) 150mg administered intramuscularly (IM) as a single-dose.
  Interventions: Drug: depo-medroxyprogesterone acetate

INTERVENTIONS:
Drug: depo-medroxyprogesterone acetate — At study entry/ Day 0, participants will receive Depo-medroxyprogesterone (DMPA) 150mg administered intramuscularly (IM) as a single-dose.
  Other Names: DMPA; Depo-Provera

SUMMARY:
This study was done to look at the level of Depo-Provera, an injectable birth control, in the blood to see whether it is affected by the anti-HIV drug Kaletra (lopinavir/ritonavir [LPV/r]). It is not known whether taking Depo-Provera together with Kaletra changes the amount of Kaletra in blood. Therefore, this study also looked at the levels of HIV and Kaletra before and after receiving a shot of Depo-Provera. This study evaluated the safety of Depo-Provera and Kaletra when they are used together. In addition to what is stated above, this study also explored any effect of Depo-Provera on the immune system.

DETAILED DESCRIPTION:
The primary study objective was addressed by calculating the Area Under the Concentration-Time Curve (AUC) from week 0 (prior to DMPA injection) to week 12 (twelve weeks after DMPA injection) in our study participants.

DMPA was supplied and administered as part of the protocol, however Kaletra was not. It was required that participants already be on a Kaletra based regimen prior to entering the study, as described in the eligibility criteria.

Arm A of AIDS Clinical Trial Group (ACTG) A5093, which consisted of 14 participants who were administered DMPA without Kaletra, was used as reference data.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Documentation of plasma HIV-1 RNA </= 400 copies/mL within 30 days prior to study entry.
* Last menstrual period </= 35 days prior to study entry.
* If last menstrual period >35 days prior to study entry, serum follicle-stimulating hormone (FSH) must be </= 40 Milli-International units per Milliliter (MIU/mL)
* Stable anti-retroviral (ARV) regimen consisting of BID LPV/r plus 2 or more nucleoside reverse transcriptase inhibitors (NRTIs) for at least 30 days if postpartum or for at least the previous 14 days if on a previously stable antiretroviral regimen without modifications prior to study entry
* Cluster of Differentiation 4 (CD4+) cell count ≥200 cells/mm^3 within 30 days prior to study entry
* Certain laboratory values within 30 days prior to study entry
* Premenopausal females with normal ovarian function
* Negative serum or urine-Human Chorionic Gonadotropin (HCG) pregnancy test within 72 hours prior to study entry
* All subjects must agree not to participate in a conception process (e.g., active attempt to become pregnant or in vitro fertilization) for the duration of the study.Subjects of reproductive potential, who are participating in sexual activity that could lead to pregnancy, must agree to use an additional reliable method of contraception while in the study.
* Ability and willingness to give written informed consent
* Documentation of Pap smear within one year prior to study entry.
* Documentation of hepatitis B (surface antigen) and hepatitis B (core antibody) and hepatitis C (antibody) status prior to study entry.
* Documentation of varicella-zoster virus (VZV) status by history of varicella or herpes zoster, or history of varicella or herpes zoster vaccination or documentation of anti-VZV antibodies.
* Willingness to abstain from alcohol 24 hours prior to and during the 10-hour pharmacokinetic (PK) specimen draws.
* Willingness to abstain from any grapefruit product or supplement for 24 hours prior to entry and for the duration of the study.

Exclusion Criteria:

* Received DMPA within 180 days prior to study entry.
* Received other hormonal therapies within the 30 days prior to study entry.
* Concurrent dual nucleoside therapy of zidovudine (ZDV) and stavudine (d4T) within 30 days prior to study entry.
* Use of any prohibited medications within 30 days prior to study entry. Prohibited Medications were:

  * amiodarone (Cordarone)
  * astemizole (Hismanal)
  * bepridil (Vascor)
  * carbamazepine (Tegretol)
  * cisapride (Propulsid)
  * clarithromycin (Biaxin)
  * cyclosporine (Sandimmune, Neoral)
  * dihydroergotamine (Migranal and others)
  * ergotamine (Ergostat, Gotamine, and others)
  * erythromycin (E-mycin, erythromycin ethylsuccinate (EES) and others)
  * flecainide (Tambocor)
  * glucocorticoids
  * Hypericum perforatum (St. John's wort)
  * itraconazole (Sporanox)
  * ketoconazole (Nizoral)
  * lovastatin (Mevacor)
  * midazolam (Versed)
  * nefazadone (Serzone)
  * phenobarbital (Luminal)
  * phenytoin (Dilantin)
  * pimozide (Orap)
  * pioglitazone (Actos)
  * propafenone (Rythmol)
  * propofol (Diprivan)
  * quinidine (Quinidex)
  * rifabutin (Mycobutin)
  * rifampin (Rifadin, Rifamate, Rifater, Rimactane)
  * rosiglitazone (Avandia)
  * simvastatin (Zocor)
  * tacrolimus (Prograf)
  * terfenadine
  * ticlopidine (Ticlid), and
  * triazolam (Halcion)
* Breastfeeding.
* Less than 30 days postpartum at study entry.
* Bilateral oophorectomy.
* Hypersensitivity to DMPA, MPA, or any of the other ingredients in DMPA.
* More than a 50% change in tobacco smoking within the 30 days prior to study entry or plans to significantly change tobacco use during the study.
* Invasive cancer of the reproductive tract; known or suspected malignancy of the breast, or known increased risk for breast cancer; undiagnosed vaginal bleeding; liver tumors; or serious ocular disorders at any time prior to study entry.
* Uncontrolled hypothyroidism or hyperthyroidism within 30 days of study entry.
* Acute infections or other opportunistic diseases requiring medication within 14 days prior to study entry.
* Receipt of any immunizations within 2 weeks prior to enrollment.
* Use of any immunosuppressant medication including systemic corticosteroids within 30 days prior to study entry.
* Chronic immunosuppressive conditions other than HIV.
* Initiated, discontinued, or changed doses of drugs that are cytochrome P450 3A4 (CYP3A4) substrates within 30 days of study entry.
* History of deep venous thrombosis or pulmonary emboli.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Cohn, M.D., M.P.H., Study Chair — Northwestern University CRS; Amneris E Luque, M.D., Study Chair — University of Rochester ACTG CRS
Locations (14):
- United States (13):
  - University of Southern California LA (5048), Los Angeles, California
  - Children's National Medical Center Washington DC NICHD CRS (5015), Washington D.C., District of Columbia
  - Washington Hospital Center NICHD CRS (5023), Washington D.C., District of Columbia
  - South Florida Childrens Diagnostic & Treatment Cen (5055), Fort Lauderdale, Florida
  - Northwestern University CRS (2701), Chicago, Illinois
  - Rush University Cook County Hospital Chicago NICHD CRS (5083), Chicago, Illinois
  - Tulane University New Orleans NICHD CRS (5095), New Orleans, Louisiana
  - Univ. of Rochester ACTG CRS (1101), Rochester, New York
  - SUNY Stony Brook NICHD CRS (5040), Stony Brook, New York
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Univ. of Cincinnati CRS (2401), Cincinnati, Ohio
  - University of Washington AIDS CRS (1401), Seattle, Washington
- San Juan Hospital PR NICHD CRS (5031), San Juan, Puerto Rico

REFERENCES:
- [Background] The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009)
- [Result] Luque AE, Cohn SE, Park JG, Cramer Y, Weinberg A, Livingston E, Klingman KL, Aweeka F, Watts DH. Depot medroxyprogesterone acetate in combination with a twice-daily lopinavir-ritonavir-based regimen in HIV-infected women showed effective contraception and a lack of clinically significant interactions, with good safety and tolerability: results of the ACTG 5283 study. Antimicrob Agents Chemother. 2015 Apr;59(4):2094-101. doi: 10.1128/AAC.04701-14. Epub 2015 Jan 26. PMID 25624326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-five HIV-1 infected women, ages 15 to 47 years, were recruited at 13 U.S. Clinical Research Sites and U.S. National Institute of Allergy and Infectious Diseases and National Institute of Child Health and Human Development-funded International Maternal Pediatric Adolescent AIDS Clinical Trial sites between June 1, 2011 and July 26, 2012.
Pre-assignment Details: Eligible participants: pre-menopausal HIV-1 infected females, >=13 years, plasma HIV-1 RNA <=400 copies/mL and cluster of differentiation 4 (CD4+) count >= 200 cells/mm^3 within 30 days prior to entry. Last menstrual period <=35 days prior to entry. If >35 days, follicle stimulating hormone (FSH) must have been <=40 Milli-International units/mL.
Groups:
- Depo-medroxyprogesterone Acetate (DMPA): At study entry/ Day 0, subjects will receive depo-medroxyprogesterone (DMPA) 150mg administered intramuscularly (IM) as a single-dose.
  depo-medroxyprogesterone acetate: At study entry/ Day 0, participants will receive Depo-medroxyprogesterone (DMPA) 150mg administered intramuscularly (IM) as a single-dose.
  Depo-medroxyprogesterone Acetate
Period: Overall Study
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Started | 25
Completed | 24
Not Completed | 1
Not completed — Unwilling to adhere to study requirement | 1

BASELINE CHARACTERISTICS:
Population: All participants enrolled.
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 22
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 31 [15 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White Non-Hispanic | 3
  Black Non-Hispanic | 15
  Hispanic (Regardless of Race) | 6
  American Indian, Alaskan Native | 1
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Medroxyprogesterone Acetate (MPA) Pharmacokinetic Parameter (PK) Area Under the Concentration-time Curve (AUC0-12weeks)
Description: This evaluates the effect of lopinavir/ritonavir (LPV/r) on pharmacokinetic parameter AUC of MPA by looking at the MPA AUC from day 0 to week 12. AUC0-12weeks was calculated using single MPA concentrations sampled immediately prior to DMPA administration on day 0, and at 2, 4, 6, 8, 10 and 12 weeks after administration of the single DMPA dose.
Time Frame: Day 0, Weeks 2, 4, 6, 8, 10 and 12
Population: One participant was excluded from all PK analyses for taking a prohibited medication with potential to interfere with PK assessments. For another participant who missed week 10 and 12 visits, a modelling approach was used to estimate the week 12 MPA level.
Measure: Median (Full Range); unit: ng*wk/mL
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
ng*wk/mL | 18.08 [5.91 to 32.33]

2. Primary Outcome: AUC0-12hour for LPV at Baseline (Day 0) Before DMPA Administration and at Week 4 (Four Weeks After DMPA Administration)
Description: This evaluates the effect of DMPA on LPV PK parameter AUC by comparing PK AUCs of LPV from 0 to 12 hours obtained at study Day 0 (before DMPA was administered) with PK AUCs of LPV from 0 to 12 hours at study Week 4 (4 weeks after DMPA was administered). Blood samples were drawn for LPV concentration levels at time zero (before LPV/r dosing) and at 30 minutes and 1, 2, 3, 4, 5, 6, 8 and 10 hours after LPV/r dosing at day 0 and week 4.
Time Frame: Day 0 and Week 4
Population: All participants eligible for the first primary PK outcome measure (MPA AUC0-12weeks) were included in this second primary outcome measure looking at LPV AUC0-12hours at Day 0 and week 4.
Measure: Median (Full Range); unit: ng*h/mL
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
ng*h/mL
  LPV AUC0-12hour at day 0 (without DMPA) | 98046.46 [38347.88 to 158899.17]
  LPV AUC0-12hour at week 4 (with DMPA) | 97948.29 [56489.42 to 192989.17]

3. Secondary Outcome: Percentage of Participants With Progesterone Levels Less Than the Lower Limit of Quantification (LLQ).
Description: This evaluates the suppression of ovulation due to the potential PK interaction between DMPA and LPV/r. The LLQ of progesterone is 0.5ng/mL. The threshold for suppression of ovulation is 5ng/mL.
Time Frame: 0, 2, 4, 6, 8, 10, and 12 weeks
Population: All 24 participants included in the primary analyses were eligible for this secondary objective, however participants occasionally missed the progesterone draw (see N for each week in table below).
Measure: Number; unit: Percent of Participants
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
Percent of Participants
  Pct with Progesterone<LLQ at Week 0 (N=24) | 50.0
  Pct with Progesterone<LLQ at Week 2 (N=23) | 87.0
  Pct with Progesterone<LLQ at Week 4 (N=24) | 95.8
  Pct with Progesterone<LLQ at Week 6 (N=24) | 95.8
  Pct with Progesterone<LLQ at Week 8 (N=24) | 95.8
  Pct with Progesterone<LLQ at Week 10 (N=20) | 95.0
  Pct with Progesterone<LLQ at Week 12 (N=23) | 95.7

4. Secondary Outcome: MPA PK Parameter Minimum Plasma Concentration (Cmin) Determined Based on MPA Levels.
Description: This evaluates the effect of LPV/r on the secondary MPA PK parameter Cmin based on MPA levels measured at weeks 0, 2, 4, 6, 8, 10, and 12.
Time Frame: 0, 2, 4, 6, 8, 10, and 12 weeks
Population: The analysis population is the 24 A5283 participants who took DMPA with LPV/r and were eligible for the primary PK outcome of MPA AUC.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
ng/mL | 0.47 [0.03 to 1.43]

5. Secondary Outcome: MPA PK Parameter Maximum Plasma Concentration (Cmax) Determined Based on MPA Levels.
Description: This evaluates the effect of LPV/r on the secondary MPA PK parameter Cmax based on MPA levels measured at weeks 0, 2, 4, 6, 8, 10, and 12.
Time Frame: 0, 2, 4, 6, 8, 10, and 12 weeks
Population: as for outcome 4
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
ng/mL | 2.88 [0.84 to 5.88]

6. Secondary Outcome: MPA PK Parameter Time to Cmax (Tmax) Determined Based on MPA Levels.
Description: This evaluates the effect of LPV/r on the secondary MPA PK parameter Tmax based on MPA levels measured at weeks 0, 2, 4, 6, 8, 10, and 12.
Time Frame: 0, 2, 4, 6, 8, 10, and 12 weeks
Population: as for outcome 4
Measure: Median (Full Range); unit: week
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
week | 4.00 [2.00 to 12.00]

7. Secondary Outcome: MPA PK Parameter Clearance (CL/F) Determined Based on MPA Levels.
Description: This evaluates the effect of LPV/r on the secondary MPA PK parameter CL/F based on MPA levels measured at weeks 0, 2, 4, 6, 8, 10, and 12.
Time Frame: 0, 2, 4, 6, 8, 10, and 12 weeks
Population: as for outcome 4
Measure: Median (Full Range); unit: L/week
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
L/week | 8297.35 [4639.14 to 25385.74]

8. Secondary Outcome: MPA PK Parameter Half-Life (T1/2) Determined Based on MPA Levels.
Description: This evaluates the effect of LPV/r on the secondary MPA PK parameter T1/2 based on MPA levels measured at weeks 0, 2, 4, 6, 8, 10, and 12.
Time Frame: 0, 2, 4, 6, 8, 10, and 12 weeks
Population: The analysis population is the 24 A5283 participants who took DMPA with LPV/r and were eligible for the primary PK outcome of MPA AUC. A minimum of three observations in the elimination phase was required to determine T1/2 and therefore results are presented for 22 participants.
Measure: Median (Full Range); unit: week
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 22
week | 3.37 [1.11 to 508.53]

9. Secondary Outcome: LPV PK Parameter Cmin.
Description: This evaluates the effect of MPA on the secondary LPV PK parameter Cmin obtained from both sampling periods, before DMPA injection at study day 0 and four weeks after DMPA injection at study week 4.
Time Frame: Day 0 and Week 4
Population: The analysis population is the 24 A5283 participants who took DMPA with LPV/r and were eligible for the primary PK outcome of LPV AUC.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
ng/mL
  LPV Cmin day 0 | 5630.00 [25.00 to 10600.00]
  LPV Cmin week 4 | 5700.00 [3630.00 to 13900.00]

10. Secondary Outcome: LPV PK Parameter Cmax.
Description: This evaluates the effect of MPA on the secondary LPV PK parameter Cmax obtained from both sampling periods, before DMPA injection at study day 0 and four weeks after DMPA injection at study week 4.
Time Frame: Day 0 and Week 4
Population: as for outcome 9
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
ng/mL
  LPV Cmax day 0 | 10750.00 [4760.00 to 16000.00]
  LPV Cmax week 4 | 10950.00 [6290.00 to 18700.00]

11. Secondary Outcome: LPV PK Parameter Tmax.
Description: This evaluates the effect of MPA on the secondary LPV PK parameter Tmax obtained from both sampling periods, before DMPA injection at study day 0 and four weeks after DMPA injection at study week 4.
Time Frame: Day 0 and Week 4
Population: as for outcome 9
Measure: Median (Full Range); unit: hour
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
hour
  LPV Tmax day 0 | 3.00 [1.00 to 8.00]
  LPV Tmax week 4 | 3.00 [1.00 to 8.00]

12. Secondary Outcome: LPV PK Parameter CL/F.
Description: This evaluates the effect of MPA on the secondary LPV PK parameter CL/F obtained from both sampling periods, before DMPA injection at study day 0 and four weeks after DMPA injection at study week 4.
Time Frame: Day 0 and Week 4
Population: as for outcome 9
Measure: Median (Full Range); unit: L/hour
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
L/hour
  LPV CL/F day 0 | 4.08 [2.52 to 10.43]
  LPV CL/F week 4 | 4.08 [2.02 to 7.08]

13. Secondary Outcome: LPV PK Parameter T1/2.
Description: This evaluates the effect of MPA on the secondary LPV PK parameter T1/2 obtained from both sampling periods, before DMPA injection at study day 0 and four weeks after DMPA injection at study week 4.
Time Frame: Day 0 and Week 4
Population: as for outcome 9
Measure: Median (Full Range); unit: hour
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
hour
  LPV T1/2 day 0 | 11.76 [1.60 to 33.67]
  LPV T1/2 week 4 | 12.64 [5.15 to 63.98]

14. Secondary Outcome: Ritonavir (RTV) PK Parameter AUC0-12h.
Description: This evaluates the effect of MPA on the PK parameter AUC0-12h of RTV obtained from both sampling periods, before DMPA injection at study day 0 and after DMPA injection at study week 4. Blood samples were drawn for RTV concentration levels at time zero (before LPV/r dosing) and at 30 minutes and 1, 2, 3, 4, 5, 6, 8 and 10 hours after LPV/r dosing at day 0 and week 4.
Time Frame: Day 0 and Week 4
Population: The analysis population is the 24 A5283 participants eligible for the primary PK outcome of LPV AUC.
Measure: Median (Full Range); unit: ng*h/mL
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
ng*h/mL
  RTV AUC0-12h day 0 | 5176.79 [1605.05 to 9858.86]
  RTV AUC0-12h week 4 | 5014.73 [2325.59 to 10011.32]

15. Secondary Outcome: RTV PK Parameter Cmin.
Description: This evaluates the effect of MPA on the PK parameter Cmin of RTV obtained from both sampling periods, before DMPA injection at study day 0 and after DMPA injection at study week 4.
Time Frame: Day 0 and Week 4
Population: The analysis population is the 24 A5283 participants eligible for the primary PK outcome of LPV AUC.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
ng/mL
  RTV Cmin day 0 | 181.00 [25.00 to 527.00]
  RTV Cmin week 4 | 194.50 [68.90 to 486.00]

16. Secondary Outcome: RTV PK Parameter Cmax.
Description: This evaluates the effect of MPA on the PK parameter Cmax of RTV obtained from both sampling periods, before DMPA injection at study day 0 and after DMPA injection at study week 4.
Time Frame: Day 0 and Week 4
Population: The analysis population is the 24 A5283 participants eligible for the primary PK outcome of LPV AUC.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
ng/mL
  RTV Cmax day 0 | 884.00 [224.00 to 2070.00]
  RTV Cmax week 4 | 726.00 [268.00 to 1950.00]

17. Secondary Outcome: RTV PK Parameter Tmax.
Description: This evaluates the effect of MPA on the PK parameter Tmax of RTV obtained from both sampling periods, before DMPA injection at study day 0 and after DMPA injection at study week 4.
Time Frame: Day 0 and Week 4
Population: The analysis population is the 24 A5283 participants eligible for the primary PK outcome of LPV AUC.
Measure: Median (Full Range); unit: hour
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
hour
  RTV Tmax day 0 | 3.00 [1.00 to 12.00]
  RTV Tmax week 4 | 3.00 [1.00 to 6.00]

18. Secondary Outcome: RTV PK Parameter CL/F.
Description: This evaluates the effect of MPA on the PK parameter CL/F of RTV obtained from both sampling periods, before DMPA injection at study day 0 and after DMPA injection at study week 4.
Time Frame: Day 0 and Week 4
Population: The analysis population is the 24 A5283 participants eligible for the primary PK outcome of LPV AUC.
Measure: Median (Full Range); unit: L/hour
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
L/hour
  RTV CL/F day 0 | 19.32 [10.14 to 62.30]
  RTV CL/F week 4 | 19.94 [9.99 to 43.00]

19. Secondary Outcome: RTV PK Parameter T1/2.
Description: This evaluates the effect of MPA on the PK parameter T1/2 of RTV obtained from both sampling periods, before DMPA injection at study day 0 and after DMPA injection at study week 4.
Time Frame: Day 0 and Week 4
Population: The analysis population is the 24 A5283 participants eligible for the primary PK outcome of LPV AUC. For one participant at day 0, T1/2 results were not estimated.
Measure: Median (Full Range); unit: hour
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
hour
  RTV T1/2 day 0 (N=23) | 4.56 [1.28 to 22.59]
  RTV T1/2 week 4 | 6.32 [2.23 to 10.62]

20. Secondary Outcome: Percentage of Participants With Menstrual Irregularities of Grade 1 and Higher Deemed Possibly, Probably or Definitely Related to Study Treatment.
Description: This evaluates toxicity and safety of concomitant medication of DMPA and LPV/r, focusing specifically on the adverse event (AE) menstrual irregularities with abnormal vaginal bleeding. The AEs were graded by the clinicians according to the Division of AIDS (DAIDS) AE Grading Table (see references in the Protocol Section) as follows: Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Potentially Life-Threatening, Grade 5=Death. Relationship to study treatment was determined by the study's co-chairs.
Time Frame: From day 0 to week 12
Population: This analysis focuses on the 24 participants eligible for the PK analyses.
Measure: Number; unit: Percent of Participants
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
Percent of Participants | 25

21. Secondary Outcome: Percentage of Participants With HIV-1 RNA Levels <400 Copies/mL.
Description: This evaluates the short-term impact of MPA on virologic suppression in participants taking LPV/r who have received a dose of DMPA by measuring percentage of participants with HIV-1 RNA levels <400 copies/mL at day 0 (prior to DMPA injection) and at weeks 2, 4, 8 and 12 (after DMPA injection). An FDA-approved HIV-1 RNA assay with a lower limit of detection of 75 copies/mL or less was required and the same HIV-1 RNA assay was required to be performed for each participant across all study visits. The Roche COBAS AmpliPrep/TaqMan HIV-1 and Abbott RealTime HIV-1 tests were used.
Time Frame: Day 0, Weeks 2, 4, 8, and 12
Population: All 24 participants included in the primary analyses were eligible for this secondary objective, however participants occasionally missed the HIV-1 RNA draw (see N for each week in table below).
Measure: Number; unit: Percent of Participants
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 24
Percent of Participants
  Pct with HIV RNA<400 at Week 0 (N=24) | 100
  Pct with HIV RNA<400 at Week 2 (N=24) | 100
  Pct with HIV RNA<400 at Week 4 (N=23) | 100
  Pct with HIV RNA<400 at Week 8 (N=24) | 100
  Pct with HIV RNA<400 at Week 12 (N=23) | 87

22. Secondary Outcome: Cell Mediated Immunity (CMI) to HIV and the Common Opportunistic Agent Varicella-zoster Virus (VZV) Using the Enzyme-linked Immunospot (ELISPOT) Assay.
Description: This evaluates the effect of MPA on CMI to HIV and VZV at baseline before DMPA (day 0) and after DMPA (weeks 4 and 12) . Cytokines are interferon-gamma (IFN-gamma) and interleukin 2 (IL-2), and Stimuli are HIV and VZV. Summary of adjusted ELISPOT assay results is in spot forming cells (SFC)/10^6 peripheral blood mononuclear cells (PBMC) by study weeks 0, 4 and 12. The outcome measures of IFN-gamma and IL-2 measured for HIV and VZV are presented here together to provide all results pertaining to the same objective in a single data table.
Time Frame: Day 0, Weeks 4 and 12
Population: All 24 participants included in the primary analyses were eligible for this secondary objective. 22 participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: SFC/10^6 PBMC
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 22
SFC/10^6 PBMC
  IFN-gamma*HIV Week 0 (N=22) | 82.50 [4.00 to 152.00]
  IFN-gamma*HIV Week 4 (N=21) | 46.50 [13.00 to 130.50]
  IFN-gamma*HIV Week 12 (N=20) | 57.75 [3.75 to 156.50]
  IFN-gamma*VZV Week 0 (N=20) | 2.75 [1.00 to 12.00]
  IFN-gamma*VZV Week 4 (N=20) | 2.00 [1.00 to 13.25]
  IFN-gamma*VZV Week 12 (N=19) | 6.50 [1.00 to 19.50]
  IL-2*HIV Week 0 (N=22) | 5.00 [1.00 to 11.50]
  IL-2*HIV Week 4 (N=21) | 4.50 [2.00 to 21.00]
  IL-2*HIV Week 12 (N=20) | 1.75 [1.00 to 5.50]
  IL-2*VZV Week 0 (N=20) | 3.25 [1.00 to 16.25]
  IL-2*VZV Week 4 (N=20) | 2.50 [1.00 to 10.00]
  IL-2*VZV Week 12 (N=19) | 5.50 [1.00 to 21.50]

23. Secondary Outcome: CMI to HIV and the Common Opportunistic Agent VZV Using the Lymphocyte Proliferation Assay (LPA).
Description: This evaluates the effect of MPA on CMI to HIV and VZV. This outcome was measured at Baseline Before DMPA (Day 0) and After DMPA (Weeks 4 and 12) using the Lymphocyte Proliferation Assay (LPA). The data table shows a summary of LPA assay results by study week with stimuli HIV and VZV. Proliferation results are reported as a stimulation index (SI) which represents the ratio of the stimulated counts per minute to unstimulated control counts per minute.
Time Frame: Day 0, Weeks 4 and 12
Population: as for outcome 22
Measure: Median (Inter-Quartile Range); unit: SI Ratio
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 22
SI Ratio
  HIV SI Week 0 (N=18) | 50.62 [5.36 to 74.13]
  HIV SI Week 4 (N=17) | 21.39 [6.99 to 50.51]
  HIV SI Week 12 (N=14) | 54.66 [5.24 to 121.13]
  VZV SI Week 0 (N=22) | 22.38 [3.05 to 66.98]
  VZV SI Week 4 (N=22) | 17.73 [4.55 to 115.22]
  VZV SI Week 12 (N=21) | 23.28 [5.02 to 148.86]

24. Secondary Outcome: Regulatory T Cells (Tregs) at Baseline, Week 4 and Week 12 Using Flow Cytometry in Freshly Thawed PBMCs.
Description: This evaluates the effect of MPA on Tregs at baseline (Day 0), week 4 and week 12 using flow cytometry in freshly thawed PBMCs. A summary of CD4+ and cluster of differentiation 8 (CD8+) anchored T-cell subsets by study week, in percent that express the marker of interest, is presented here together to provide all results pertaining to this objective in a single data table.
Time Frame: Day 0, Weeks 4 and 12
Population: All 24 participants included in the primary analyses were eligible for this secondary objective. 21 participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: Percent CD4/CD8 cells expressing marker
Arm/Group | Depo-medroxyprogesterone Acetate (DMPA)
Number analyzed (Participants) | 21
Percent CD4/CD8 cells expressing marker
  CD4+FOXP3+ Week 0 | 1.26 [0.80 to 2.73]
  CD4+FOXP3+ Week 4 | 1.30 [0.90 to 1.46]
  CD4+FOXP3+ Week 12 | 1.29 [1.01 to 1.80]
  CD4+CD25+FOXP3+ Week 0 | 0.41 [0.17 to 0.80]
  CD4+CD25+FOXP3+ Week 4 | 0.24 [0.11 to 0.62]
  CD4+CD25+FOXP3+ Week 12 | 0.33 [0.13 to 0.45]
  CD4+CD39+ Week 0 | 10.10 [5.95 to 15.90]
  CD4+CD39+ Week 4 | 10.10 [6.31 to 13.20]
  CD4+CD39+ Week 12 | 11.60 [7.65 to 16.50]
  CD4+TGFB+ Week 0 | 4.32 [2.66 to 6.02]
  CD4+TGFB+ Week 4 | 3.62 [1.93 to 7.96]
  CD4+TGFB+ Week 12 | 3.08 [2.30 to 5.62]
  CD4+IL10+ Week 0 | 4.66 [3.52 to 6.16]
  CD4+IL10+ Week 4 | 6.01 [3.41 to 7.68]
  CD4+IL10+ Week 12 | 5.64 [3.56 to 8.43]
  CD4+IL35+ Week 0 | 1.86 [1.22 to 3.36]
  CD4+Interleukin35+(IL35+) Week 4 | 1.59 [0.93 to 3.19]
  CD4+IL35+ Week 12 | 1.35 [0.78 to 2.08]
  CD8+FOXP3+ Week 0 | 0.85 [0.54 to 1.04]
  CD8+FOXP3+ Week 4 | 0.91 [0.68 to 1.49]
  CD8+FOXP3+ Week 12 | 0.74 [0.67 to 1.43]
  CD8+CD25+FOXP3+ Week 0 | 0.07 [0.03 to 0.19]
  CD8+CD25+FOXP3+ Week 4 | 0.06 [0.03 to 0.27]
  CD8+CD25+FOXP3+ Week 12 | 0.08 [0.01 to 0.26]
  CD8+CD39+ Week 0 | 3.38 [2.53 to 4.52]
  CD8+CD39+ Week 4 | 4.20 [2.37 to 4.89]
  CD8+CD39+ Week 12 | 3.12 [2.31 to 5.20]
  CD8+TGFB+ Week 0 | 1.26 [0.74 to 1.90]
  CD8+TGFB+ Week 4 | 1.22 [0.76 to 2.02]
  CD8+TGFB+ Week 12 | 1.18 [0.60 to 1.66]
  CD8+IL10+ Week 0 | 1.46 [1.10 to 1.87]
  CD8+IL10+ Week 4 | 1.53 [1.13 to 2.60]
  CD8+IL10+ Week 12 | 1.45 [1.10 to 2.21]
  CD8+IL35+ Week 0 | 1.22 [0.87 to 1.61]
  CD8+IL35+ Week 4 | 1.52 [0.53 to 1.99]
  CD8+IL35+ Week 12 | 0.89 [0.65 to 1.83]

ADVERSE EVENTS:
Time Frame: From Day 0 to Week 12.
Description: The serious adverse event (SAE) Reporting Category, as defined in Version 2.0 of the DAIDS expedited adverse events (EAE) Manual was used for this study. Study agents requiring expedited reporting were: DMPA and LPV/r.
  The DAIDS AE Grading Table, Version 1.0, December 2004 (Clarification, August 2009) was used to grade the severity of events.
Groups:
- Arm A: At study entry/ Day 0, subjects will receive depo-medroxyprogesterone (DMPA) 150mg administered intramuscularly (IM) as a single-dose.
Arm/Group | Arm A
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 9/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=25)
Chills (General disorders) | 2
Weight increased (Investigations) | 2
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Irritability (Psychiatric disorders) | 2
Menorrhagia (Reproductive system and breast disorders) | 4
Metrorrhagia (Reproductive system and breast disorders) | 5
Vaginal haemorrhage (Reproductive system and breast disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No